CLINICAL TRIAL: NCT05117593
Title: Phase 1 Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single-Ascending Doses of FBL-MTX in Healthy Subjects
Brief Title: Investigate the Safety, Tolerability and Pharmacokinetics of FBL-MTX
Acronym: FolSmart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SOLFARCOS - Pharmaceutical and Cosmetic Solutions Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: FBL-MTX-101
Record Dates: First submitted 2021-09-23; First posted 2021-11-11 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; healthy
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: A maximum of 4 dose levels (0.1 mg, 0.33 mg, 1 mg and 2.5 mg) is preplanned to be investigated in separate sequential cohorts. Each cohort will consist of 8 healthy male and female subjects (3 subjects of either sex on FBL-MTX, 1 of either sex on placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBL-MTX (Experimental): A single dose of FBL-MTX will be administered by slow intravenous injection in the morning, under fasted conditions.
  A maximum of 4 dose levels (0.1 mg, 0.33 mg, 1 mg and 2.5 mg) are pre-planned.
  Interventions: Drug: FBL-MTX
- Placebo (Placebo Comparator): A single dose of placebo will be administered by slow injection in the morning, under fasted conditions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FBL-MTX — FBL-MTX is available as sterile liposomal dispersion for injection at nominal dose strength of 1 mg/mL of methotrexate free base. The dose of 0.1 mg was selected as starting dose in the present study. Three subsequent FBL-MTX dose levels are pre-planned: 0.33 mg, 1 mg and 2.5 mg.
  Arms: FBL-MTX
Drug: Placebo — Placebo will consist of sterile saline 0.9% NaCl solution.
  Arms: Placebo

SUMMARY:
This is a prospective, single-center, randomized, double-blind, placebo-controlled, single-ascending dose (SAD) phase 1 study to evaluate the safety, tolerability and pharmacokinetics of FBL-MTX in healthy male and female subjects.

DETAILED DESCRIPTION:
The product FBL-MTX consists of Methotrexate (MTX) encapsulating liposomes functionalized with a folate peptide (SP-DS3), which targets activated macrophages of rheumatoid arthritis (RA).

This is a prospective, single-center, randomized, double-blind, placebo-controlled, single-ascending dose (SAD) phase 1 study in healthy subjects.

This study is planned to investigate up to 4 dose levels of FBL-MTX. Each dose level will consist of 8 healthy male and female subjects (ratio 1:1, male:female) to have 6 subjects being administered FBL-MTX and 2 subjects being administered placebo (ratio 3:1, active:placebo).

The study is designed to meet the following objectives:

* Primary: To evaluate the safety and tolerability of FBL-MTX following single-ascending intravenous doses to healthy male and female subjects.
* Secondary: To investigate the PK of FBL-MTX following single-ascending intravenous doses to healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-mandated procedure.
2. Healthy male or female subjects aged between 18 and 55 years (inclusive) at Screening.
3. Body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive) at Screening.
4. Ability to communicate well with the investigator, in a language understandable to the subject, and to understand and comply with the study requirements.
5. Systolic blood pressure (SBP) 100-140 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and pulse rate 50-90 bpm (inclusive), measured on the same arm after ≥5 min in the supine position, at Screening and on Day -1.
6. Estimated glomerular filtration rate calculated using the Cockcroft-Gault equation ≥ 90 mL/min at Screening.
7. A female subject of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1 and must agree to consistently and correctly use (from Screening, during the entire study, and for at least 6 months after investigational product administration) a highly effective method of contraception with a failure rate of ≤1% per year, be sexually inactive, or have a vasectomized partner. If a hormonal contraceptive is used, it must be initiated at least 1 month before the treatment administration.
8. A female subject of non-childbearing potential, must be post-menopausal (defined as 12 consecutive months with no menses without an alternative medical cause, confirmed by a follicle stimulating hormone [FSH] test), or must have a medical history of previous bilateral salpingectomy, bilateral salpingo-oophorectomy, hysterectomy, premature ovarian failure (confirmed by a specialist), XY genotype, Turner syndrome, or uterine agenesis.
9. A male subject must use adequate contraception (e.g., condom) from investigational product administration up to at least 6 months after, unless he is vasectomized or sexually inactive. In addition, the subject must ensure that his female partner of childbearing potential agrees to consistently and correctly use for the same period a highly effective method of contraception with a failure rate of ≤1% per year.
10. A male subject must agree to refrain from donation of semen from investigational product administration up to at least 6 months after.

Exclusion Criteria:

1. Previous exposure to FBL-MTX.
2. Known hypersensitivity to MTX or any other FBL-MTX components.
3. Clinically relevant findings on physical examination at Screening or on Day -1.
4. Clinically relevant abnormalities on 12-lead ECG, measured after 5 min in a supine position, at Screening or on Day -1.
5. Clinically relevant abnormalities on chest X-ray at Screening.
6. Clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry, and urinalysis) at Screening or on Day -1.
7. Pre-existing blood dyscrasias, such as bone marrow hypoplasia, leukopenia, thrombocytopenia or significant anemia.
8. QTc > 450ms in male and > 470ms in female.
9. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) above the normal range.
10. Any medical condition, acute, ongoing, recurrent or chronic, that presents a potential risk to the participant and/or that may compromise the objectives of the study.
11. History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the distribution, metabolism, or excretion of the investigational product.
12. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator.
13. History of tuberculosis.
14. Presence of chronic or acute bacterial or viral infection.
15. History or presence of an autoimmune disorder.
16. History of known or suspected immunodeficiency syndrome
17. Stomatitis, ulcers of the oral cavity and known active gastrointestinal ulcer disease.
18. Any significant acute or chronic medical illness, including past or present liver disease.
19. Previous clinically relevant history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
20. Veins unsuitable for intravenous puncture on either arm (e.g., veins that are difficult to locate, access, or puncture, veins with a tendency to rupture during or after puncture).
21. Participation in a clinical study involving investigational product administration within 3 months prior to Screening or in more than 2 clinical studies within 1 year prior to Screening.
22. History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to Screening.
23. Excessive methylxanthines consumption, defined as ≥ 500 mg per day, at Screening.
24. Nicotine intake (e.g., smoking, nicotine patch, nicotine chewing gum, or electronic cigarettes) within 3 months prior to Screening and inability to refrain from nicotine intake from Screening up to End-of-Study (EOS).
25. Previous treatment with any prescribed medications or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 3 weeks prior to investigational product administration.
26. Previous treatment with vaccines within 4 weeks prior to investigational product administration.
27. Loss of 250 mL or more of blood within 3 months prior to Screening.
28. Positive results from urine drug and alcohol screen at Screening or on Day -1.
29. Positive Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) and/or HCV antibodies at Screening.
30. Positive HIV serology results at Screening.
31. Pregnant or lactating woman.
32. Any other circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline at each time point of measurement in systolic blood pressure | From study treatment administration up to end of study, an average of 1month
  Measurements must be recorded from the subject in the supine position after having rested for at least 5 min
Change from baseline at each time point of measurement in diastolic blood pressure | From study treatment administration up to end of study, an average of 1month
  Measurements must be recorded from the subject in the supine position after having rested for at least 5 min
Change from baseline at each time point of measurement in pulse rate | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in hemoglobin | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in red cell count | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in hematocrit | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in mean corpuscular volume | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in mean corpuscular hemoglobin | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in mean corpuscular hemoglobin concentration | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in red cell distribution width | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in white cell count with differential | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in platelet count | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in mean platelet volume | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in AST | From study treatment administration up to end of study, an average of 1 month
  Measurement of aspartate aminotransferase
Change from baseline at each time point of measurement in clinical ALT | From study treatment administration up to end of study, an average of 1 month
  Measurement of alanine aminotransferase
Change from baseline at each time point of measurement in gamma-glutamyltransferase (GGT) | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in alkaline phosphatase (ALP) | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in total bilirubin | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in indirect bilirubin | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in direct bilirubin | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in lactate dehydrogenase (LDH) | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in creatinine | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in urea | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in urate | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in glucose | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in cholesterol | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in triglycerides | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in sodium | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in potassium | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in chloride | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in calcium | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in protein | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in albumin | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in creatine kinase (CK) | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in creatinine clearance | From study treatment administration up to end of study, an average of 1 month
Change from baseline at each time point of measurement in glucose in urine | From study treatment administration up to end of study, an average of 1 month
  Urinalysis test
Change from baseline at each time point of measurement in bilirubin in urine | From study treatment administration up to end of study, an average of 1 month
  Urinalysis test
Change from baseline at each time point of measurement in ketone in urine | From study treatment administration up to end of study, an average of 1 month
  Urinalysis test
Change from baseline at each time point of measurement in specific gravity | From study treatment administration up to end of study, an average of 1 month
  Urinalysis test
Change from baseline at each time point of measurement in hemoglobin in urine | From study treatment administration up to end of study, an average of 1 month
  Urinalysis test
Change from baseline at each time point of measurement in pH in urine | From study treatment administration up to end of study, an average of 1 month
  Urinalysis test
Change from baseline at each time point of measurement in protein in urine | From study treatment administration up to end of study, an average of 1 month
  Urinalysis test
Change from baseline at each time point of measurement in urobilinogen | From study treatment administration up to end of study, an average of 1 month
  Urinalysis test
Change from baseline at each time point of measurement in nitrite in urine | From study treatment administration up to end of study, an average of 1 month
  Urinalysis test
Change from baseline at each time point of measurement in heart rate | From study treatment administration up to the end of study, an average of 1 month
Change from baseline at each time point of measurement in QT interval corrected with Bazett's formula | From study treatment administration up to the end of study, an average of 1 month
Change from baseline at each time point of measurement in QT interval corrected with Fridericia's formula (QTcF) | From study treatment administration up to the end of study, an average of 1 month
Treatment-emergent AEs | From study treatment administration up to the end of study, an average of 1 month
Treatment-emergent SAEs | From study treatment administration up to the end of study, an average of 1 month
Treatment-emergent AEs leading to premature study discontinuation. | From study treatment administration up to the end of study, an average of 1 month

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Multiple pharmacokinetic sampling at predefined timepoints from Day 1 (pre-dose) up to Day 7.
Time to reach Cmax (tmax). | Multiple pharmacokinetic sampling at predefined timepoints from Day 1 (pre-dose) up to Day 7.
  If the maximum value occurs at more than one timepoint, tmax is defined as the first time point with this value
Area under the concentration-time curve (AUC) from time zero to last measurable plasma concentration (AUC0-t) | Multiple pharmacokinetic sampling at predefined timepoints from Day 1 (pre-dose) up to Day 7.
  Calculated using the linear trapezoidal rule.
AUC from time zero to infinity (AUC0-∞) | Multiple pharmacokinetic sampling at predefined timepoints from Day 1 (pre-dose) up to Day 7.
  Calculated as follows: AUC0-∞ = AUC0-t + Ct/λz, where Ct is the last quantifiable concentration at time t and λz is the apparent terminal elimination rate constant.
Terminal elimination rate constant (λz). | Multiple pharmacokinetic sampling at predefined timepoints from Day 1 (pre-dose) up to Day 7.
Terminal elimination half-life (t1/2). | Multiple pharmacokinetic sampling at predefined timepoints from Day 1 (pre-dose) up to Day 7.
Apparent plasma clearance (CL/F). | Multiple pharmacokinetic sampling at predefined timepoints from Day 1 (pre-dose) up to Day 7.
  Calculated as Dose / AUC0-∞.
Apparent volume of distribution (Vz/F) during the terminal elimination phase | Multiple pharmacokinetic sampling at predefined timepoints from Day 1 (pre-dose) up to Day 7.
  Calculated as Dose / (AUC0-∞ . λz).

CONTACTS AND LOCATIONS:
Locations (1):
- BlueClinical Phase I, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No